CLINICAL TRIAL: NCT06369272
Title: An Observational Study to Assess Maternal and Infant Outcomes Following Exposure to SPIKEVAX During Pregnancy
Brief Title: Study to Assess Maternal and Infant Outcomes Following Exposure to SPIKEVAX During Pregnancy
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P919
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Maternal Outcomes; Infant Outcomes; Pregnancy
Keywords: Maternal outcomes; Infant outcomes; Pregnancy; Observational; SPIKEVAX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- SPIKEVAX Exposed Pregnancy: Cohort includes pregnant women who were vaccinated with SPIKEVAX from last menstrual period (LMP) through the exposure ascertainment period for the outcome of interest.
- SPIKEVAX Distantly Exposed Pregnancy: Cohort includes pregnant women who were exposed to SPIKEVAX at least 60 days prior to LMP and not exposed to SPIKEVAX or any other COVID-19 vaccine from LMP through the exposure ascertainment period for the outcome of interest.
- Unvaccinated During Pregnancy: Cohort includes pregnant women not exposed to SPIKEVAX or any other COVID-19 vaccine within 60 days prior to LMP through the exposure ascertainment period for the outcome of interest.
- COVID-19 Infected During Pregnancy: Cohort includes pregnant women not exposed to SPIKEVAX or any other COVID-19 vaccine within 60 days prior to LMP through the exposure ascertainment period for the outcome of interest. These women also had at least one medically attended COVID-19 episode during the exposure ascertainment period outcome of interest.

SUMMARY:
The primary objectives of this study are:

In infants of women exposed to SPIKEVAX during pregnancy, to assess:

* If exposure to SPIKEVAX during pregnancy is associated with an increased birth prevalence of major congenital malformations (MCMs).
* If exposure to SPIKEVAX during pregnancy is associated with an increased birth prevalence of adverse neonatal and infant outcomes, specifically neonatal encephalopathy, small for gestational age, respiratory distress in the newborn, and incidence of hospitalization due to infections including coronavirus disease 2019 (COVID-19).
* In women exposed to SPIKEVAX during pregnancy, to assess whether exposure to SPIKEVAX is associated with an increased prevalence of hypertensive disorders [e.g., pre-eclampsia, eclampsia, and gestational hypertension] gestational diabetes, and post-partum hemorrhage; and
* To assess whether exposure to SPIKEVAX during pregnancy is associated with an increased incidence of stillbirth, preterm birth, and medically attended spontaneous abortion.

ELIGIBILITY:
Inclusion Criteria:

* EOP within study period
* Continuous enrollment in a health plan contributing to the HealthCare Integrated Research Database℠ (HIRD) database for at least 90 days prior to the estimated LMP.

Exclusion Criteria:

* Exposure to any non-Moderna COVID-19 vaccines at any time prior to LMP and from LMP through the exposure ascertainment period for the outcome of interest. However, pregnant women exposed to other non-Moderna vaccines in addition to SPIKEVAX will be included in a sensitivity analysis.
* Instances where the outcome of a pregnancy is not documented (e.g., a prenatal care claim is followed by no further documentation of pregnancy, termination, or delivery where the participant remains enrolled in the health plan) may also be observed. The number of these possibly exposed pregnancies will be tabulated and described; however, they will not be included in the descriptive or comparative analyses.

Ages: 13 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population includes women for whom an LMP can be successfully calculated based on a non-missing end of pregnancy (EOP), and who also meet the eligibility criteria to be included in the study analyses.
Sampling Method: Non-Probability Sample
Enrollment: 1192 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Number of MCMs | Up to approximately 3 years
Number of Adverse Neonatal and Infant Outcomes | Up to approximately 3 years
  Adverse neonatal and infant outcomes include neonatal encephalopathy, small for gestational age, respiratory distress in the newborn, or incidence of hospitalization due to infections including COVID-19.
Number of Participants with Hypertensive Disorders | Up to approximately 3 years
  Hypertensive disorders include pre-eclampsia, eclampsia, and gestational hypertension, gestational diabetes, or post-partum hemorrhage
Number of Stillbirths, Preterm Births, and Medically Attended Spontaneous Abortions | Up to approximately 3 years

SECONDARY OUTCOMES:
Demographics: Participant Region of Residence | Baseline
Demographics: Age at LMP | Baseline
Demographics: Number of Overweight or Obese Participants | Baseline
Demographics: Duration of Health Plan Enrolment Prior to Pregnancy | Baseline
Demographics: Calendar Date of the Pregnancy Outcome | Baseline
Demographics: Participant Race and Ethnicity | Baseline
Demographics: Participant Socio-economic Status | Baseline
Healthcare Utilization: Number of Office Visits, Emergency Department Visits, and Hospitalizations | Baseline
Healthcare Utilization: Number of Distinct Medications Used | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Carelon Research, Newton, Massachusetts, United States